CLINICAL TRIAL: NCT02619773
Title: The Use of Mupirocin Dressings and Its Effect on Surgical Site Infections in Elective Colorectal Surgery: A Prospective, Randomized Controlled Trial
Brief Title: Effect of Mupirocin Dressings Versus Island Dressings on Surgical Site Infections in Elective Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Collaborators: Gundersen Lutheran Health System (Other)
Responsible Party: Principal Investigator, Kara Kallies, Academic Researcher, Gundersen Lutheran Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2-15-10-001
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Surgical Site Infections
Keywords: Colorectal Surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mupirocin dressing (Experimental): Mupirocin + island dressing applied to surgical incision until postoperative day 5.
  Intervention: mupirocin ointment applied to extrication incision.
  Interventions: Procedure: mupirocin ointment
- Island dressing (No Intervention): Island dressing applied to surgical incision until postoperative day 2. This arm will not undergo any intervention.

INTERVENTIONS:
Procedure: mupirocin ointment — Mupirocin ointment will be applied after skin closure. A standard island dressing will be placed over the incision.
  Arms: Mupirocin dressing

SUMMARY:
Infections at the site of surgical incisions (SSIs) are the most common infection among surgical patients. Although all patients undergoing surgical procedures are at risk for developing SSIs, colorectal surgery has had consistently had high rates of SSIs, ranging from 3-45%. These infections can increase the length of hospital stay, and increase the rate of readmissions and costs.

Further research is needed to study the effects of mupirocin in general surgery. A recent study compared colorectal SSI rates between mupirocin and standard gauze surgical dressings. The results of this show that mupirocin has the greatest effect on reducing SSI rate when compared to standard gauze dressings. However, these studies have not been performed in the United States and have only been studied on a very specific patient population.

The purpose of this study is to assess the rate of infections at the surgical incision after colorectal surgery when a mupirocin dressing is placed versus a standard gauze dressing without mupirocin.

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are the most common nosocomial infection among surgical patients and are the third most common nosocomial infection among all hospitalized patients.1 Although all patients undergoing surgical procedures are at risk for developing SSIs, colorectal surgery has consistently had high rates of surgical site infections, ranging from 3-45%. Numerous studies have shown the adverse effects of SSIs, including increased length of hospital stay, morbidity, mortality, readmissions and costs. In a recent study analyzing various surgical procedures, including colorectal operations, surgical site infection was found to be the number one cause of unplanned readmission.

Studies have been performed showing that intranasal mupirocin may have a role in reduction of SSI in cardiac and orthopedic surgery. However, there has been minimal investigation on the effects of topical mupirocin in general surgery. A recent study from Spain compared colorectal SSI rates between mupirocin dressings, silver-impregnated dressings, and standard gauze surgical dressings. The results of this show that mupirocin has the greatest effect on reducing SSI rate when compared to standard gauze and silver-impregnated dressings. However, these studies have not been performed in the United States and have only been studied on open, colorectal oncologic surgery.

The aim of this study is to compare mupirocin dressings to standard surgical dressings and their respective SSI rates at a United States community hospital in patients undergoing elective open and minimally invasive colorectal surgery.

A single-center prospective, randomized study will be performed. Patients who will undergo elective colorectal surgery and consent to participate will be randomized (1:1) to one of the following 2 treatment groups:

1. Island dressings until postoperative day (POD) #2 (which is current practice at Gundersen Health System)
2. Mupirocin + island dressing until POD#5 Analysis of outcomes will include rate of SSI, and 30-day morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Elective Colorectal surgery
* Open and minimally invasive cases
* Partial and total Colon resections, Abdominoperineal resection, Low anterior resections, Creation/takedown of colostomy, abdominal procedures for prolapse

Exclusion Criteria:

* Patients with known allergies to mupirocin
* Cases in which the skin was intentionally left open at the end of surgery (secondary closure technique)
* Women who are pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | within 30 days postoperative
  Surgical site infection defined per ACS NSQIP criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Shapiro, MD, Principal Investigator — Gundersen Health System
Locations (1):
- Gundersen Lutheran Health System, La Crosse, Wisconsin, United States